CLINICAL TRIAL: NCT02242240
Title: Lung Function Changes Following the Addition of Formoterol Inhalation Capsules (12 µ Once or Twice Daily) to Pharmacodynamic Steady State of Once Daily Tiotropium (18 µg) Inhalation Capsule in Patients With COPD
Brief Title: Lung Function Changes Following the Addition of Formoterol to Tiotropium in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1184.2
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (3):
- Tiotropium with single dose of formoterol (Experimental)
  Interventions: Drug: Formoterol once daily; Drug: Tiotropium once daily
- Tiotropium with double dose of formoterol (Experimental)
  Interventions: Drug: Formoterol twice daily; Drug: Tiotropium once daily
- Tiotropium with Placebo (Experimental)
  Interventions: Drug: Tiotropium once daily; Drug: Placebo

INTERVENTIONS:
Drug: Formoterol twice daily
  Arms: Tiotropium with double dose of formoterol
Drug: Formoterol once daily
  Arms: Tiotropium with single dose of formoterol
Drug: Tiotropium once daily
Drug: Placebo
  Arms: Tiotropium with Placebo

SUMMARY:
Study to establish the lung function effects of added formoterol (12μg QD and BID) during 2-week periods to pharmacodynamic steady state of tiotropium(18μg QD)

ELIGIBILITY:
Inclusion Criteria:

* All patients must sign an informed consent consistent with international conference of harmonization (ICH)-good clinical practice (GCP) guidelines prior to participation in the trial, which includes medication washout and restrictions
* All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

  * Patients must have relatively stable* moderate to severe airway obstruction with an FEV1 ≤ 60% of predicted normal and FEV1 ≤ 70% of FVC (Visit 1)

    * Patients who have frequent exacerbations (at least three in the preceding year) which could be expected to interfere with the patient's ability to participate in the trial should be excluded. The enrollment of patients who have had an exacerbation within the six-week period prior to planned study entry should be postponed for at least six weeks
  * Predicted normal values will be calculated according to european community for coal and steel (ECCS):
  * Males: FEV1 predicted (L) = 4.30 x Height (metres) - 0.029 x Age (years) - 2.49
  * Females: FEV1 predicted (L) = 3.95 x Height (metres) - 0.025 x Age (years) - 2.60
* Male or female patients 40 years of age or older
* Patients must be current or ex-smokers with a smoking history of more than 10 pack-years

  * patients who have never smoked cigarettes must be excluded
* Patients must be able to perform technically acceptable pulmonary function tests and must be able to maintain records (Patient Daily Record) during the study period as required in the protocol
* Patients must be able to inhale medication from inhalation capsule delivery systems (the HandiHaler® for the tiotropium and placebo capsules and the Aerolizer® for the formoterol capsule) and from a metered dose inhaler

Exclusion Criteria:

* Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
* Patients with clinically relevant abnormal baseline hematology, blood chemistry, or urinalysis if the abnormality defines a disease listed as an exclusion criterion
* All patients with a serum glutamate oxaloacetate transaminase (SGOT) > 80 IU/L, serum glutamate pyruvate transaminase (SGPT) > 80 IU/L, bilirubin > 17 µmol/L or creatinine > 110 µmol/L (males) / 95 µmol/L (females) will be excluded regardless of clinical condition. Repeat laboratory evaluation will not be conducted in these patients
* Patients with a recent history (i.e., six months or less) of myocardial infarction
* Patients with any cardiac arrhythmia requiring drug therapy or who have been hospitalized for heart failure within the past three years
* Patients with known active tuberculosis
* Patients on oxygen therapy
* Patients with history of cystic fibrosis, bronchiectasis, interstitial lung disease, or pulmonary thromboembolic disease
* Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion 1
* Patients with any respiratory infection in the six weeks prior to the Screening Visit (Visit 1) or during the baseline period
* Patients with known hypersensitivity to anticholinergic drugs, beta adrenergics, lactose or any other components of the inhalation capsule delivery system
* Patients with a history of cancer within the last three years. Patients with treated basal cell carcinoma are allowed. Patients with successfully treated cancers greater than five years prior to entry will be allowed
* Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction
* Patients with known narrow-angle glaucoma
* Patients using cromolyn sodium or nedocromil sodium
* Patients using treated with antihistamines (H1 receptor antagonists)
* Patients using treated with theophyllines
* Patients on ß-blocker therapy
* Patients using oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception for the previous 3 months (i.e. oral contraceptives, intrauterine devices, diaphragm or subdermal implants e.g., Norplant®)
* Patients with a history of asthma, allergic rhinitis or atopy or who have a total blood eosinophil count ≥ 600 mm3. A repeat eosinophil count will not be conducted in these patients
* Patients with significant alcohol or drug abuse within the past two years
* Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to Screening Visit (Visit 1)
* Patients who are currently in a pulmonary rehabilitation program or who have completed a program in the six weeks prior to screening (Visit 1)
* Patients who currently participating in another study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2001-03; Primary Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time point zero to 24 hours (AUC0-24h) for forced expiratory volume in one second (FEV1) | Pre-dose, up to 24 hours after start of treatment
Area under the curve from 12 to 24 hours (AUC12-24h) for forced expiratory volume in one second (FEV1) | 12 to 24 hours after start of treatment

SECONDARY OUTCOMES:
Trough FEV1 response on each pulmonary function test day | 24 hours after intake of the last morning dose
Trough forced vital capacity (FVC) response on each pulmonary function test day | Up to 24 hours after start of treatment
FEV1 AUC0-12h on each pulmonary function test day | Up to 12 hours after start of treatment
Individual FEV1measurements at each time point | up to day 58 day after start of treatment
Individual FVC measurements at each time point | up to day 58 day after start of treatment
Individual inspiratory capacity (IC) measurements at each time point | up to day 58 day after start of treatment
Peak expiratory flow rate (PEFR) measured by the patients at home twice daily | up to day 79 after start of treatment
Amount of salbutamol therapy used during the treatment period | up to day 79 after start of treatment
Number of patients with adverse events | Up to 93 days
FVC AUC0-12h on each pulmonary function test day | up to day 58 day after start of treatment
Peak FEV1 response on each pulmonary function test day | within 3 hours after treatment
Peak FVC response on each pulmonary function test day | within 3 hours after treatment